CLINICAL TRIAL: NCT07375667
Title: Mechanisms of Dynamic Airway Resistance Monitoring and Machine Learning for Assessing Pulmonary Inflammation and Guiding Sputum Suction in Mechanically Ventilated Patients
Brief Title: Dynamic Airway Resistance & ML: Guide Sputum Suction in Ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-K249-01
Record Dates: First submitted 2025-12-10; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: Mechanical Ventilation Pressure High; Ventilator-Associated Pneumonia (VAP); Respiratory Depression Neonatal
Keywords: Airway resistance
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Airway resistance-guided sputum suction (Experimental): Investigators will continuously monitor the airway viscous resistance of patients, and initiate suctioning when the airway viscous resistance increases by ≥6 cmH₂O.
  Interventions: Procedure: The dynamics of airway resistance; Diagnostic Test: conventional suctioning
- conventional suctioning (No Intervention): In the control group, the decision to suction was made based on conventional clinical signs, including rhonchi and a rise in peak pressure.

INTERVENTIONS:
Procedure: The dynamics of airway resistance — Monitoring the dynamic changes in airway resistance in patients can be used to reflect the progression of pulmonary inflammation and determine the optimal timing for suctioning.
  Arms: Airway resistance-guided sputum suction
Diagnostic Test: conventional suctioning — The timing for suctioning is determined based on clinical signs such as rhonchi and an elevated peak pressure.
  Arms: Airway resistance-guided sputum suction

SUMMARY:
Research has shown that timely suctioning not only improves survival rates but also enhances the quality of life in ventilator-dependent patients. However, clinical judgment on the optimal timing for suctioning currently relies primarily on physician experience, lacking scientific evidence [10]. Airway viscous resistance reflects the frictional resistance encountered by gas flow within the airways and is closely associated with airway patency. When airway secretions increase, viscous resistance undergoes dynamic changes. Therefore, analyzing these dynamic variations in viscous resistance derived from ventilator waveforms to determine the optimal suctioning timing and assess its clinical impact on the progression of pulmonary inflammation holds significant scientific value and offers new insights and methodologies for clinical practice.

DETAILED DESCRIPTION:
To validate the clinical feasibility and reliability of airway viscous resistance monitoring, explore the temporal correlation between inflammatory biomarkers and changes in airway viscous resistance, establish a reference threshold system for special populations, and provide experimental evidence for determining the optimal suctioning timing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute Respiratory Distress Syndrome (ARDS)
* Clinical diagnosis of Acute Exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD)
* Clinical diagnosis of Severe pneumonia

Exclusion Criteria:

* Clinical diagnosis of multiple organ failure;
* Clinical diagnosis of multiple organ bleeding;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
The drop in airway viscous resistance before and after sputum suction | the process of sputum aspiration(at most 30 minutes)
  Airway viscous resistance drop (AVRD) is the primary efficacy endpoint of this study. It is defined as the difference in airway viscous resistance measured immediately before and after suctioning.
  Procedure: Record the ventilator-displayed viscous resistance value pre-suction; immediately after the maneuver, re-measure both viscous resistance and peak airway pressure with a high-precision pressure-time sensor.
  Calculation: The within-patient difference (pre minus post) is the AVRD. In a pilot study of nine patients, AVRD averaged 6.889 ± 3.551 cmH₂O, significantly larger than the concurrent peak-pressure drop (1.556 ± 1.740 cmH₂O), indicating that AVRD is more sensitive to the effect of suction on airway secretions.
  Clinical implication: AVRD can serve as a quantitative criterion for determining the optimal timing of endotracheal suction.

SECONDARY OUTCOMES:
The number of participants with abnormal laboratory tests | Laboratory testing time ( at least 30 minutes)
  Venous blood testing was performed, including a complete blood count (white blood cell count [WBC], neutrophil percentage [NEUT%]), C-reactive protein (CRP), and procalcitonin (PCT) to assess the systemic inflammatory status.
Sputum bacterial culture | 3 days
  Sputum culture is performed to identify the source of infection and to diagnose VAP.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - the Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
All data
Supporting Information: CSR
Time Frame: From October 2025 until the end of the trial
Access Criteria: Critical care researchers; all materials will be made available. Contact: Honglei Wu, e-mail: wu_honglei@163.com
URL: https://www.ahnmc.com/